CLINICAL TRIAL: NCT05562908
Title: Skeletonised Versus Pedicled Internal Thoracic Artery - A Randomised Study
Brief Title: Skeletonised Versus Pedicled Internal Thoracic Artery
Acronym: TST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lars Peter Riber (Other)
Collaborators: Odense Patient Data Explorative Network (Other); GCP-unit at Odense University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Lars Peter Riber, MD, Associate Professor, Ph.D., DMSc, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP_764; S-20180083 (Registry Identifier: The Danish ethical committee - region of southern Denmark)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Heart Diseases
Keywords: coronary artery diseases; left internal mammary artery; LIMA harvesting; flow; quality of life
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease | interventions — Surgical Flaps

STUDY DESIGN:
Intervention Model Description: Randomised trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: After randomisation, the attending consultant informed the patient of the harvesting method. Data collector and outcome adjudicator were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pedicled (Active Comparator): Harvesting of LIMA with its surrounding tissue: fascia, veins, etc
  Interventions: Procedure: Pedicled
- Surgical skeletonised (Active Comparator): Harvesting of LIMA in a "naked" fashion where you dissect the artery free of the surrounding tissue.
  Interventions: Procedure: Surgical skeletonised
- Skeletonised with Thunderbeat (Active Comparator): Same as Surgical skeletonised but instead of closing the side branches with clips a surgical tool is used for coagulation of the side-branches.
  Interventions: Procedure: Thunderbeat skeletonised

INTERVENTIONS:
Procedure: Pedicled — Surgical procedure: A prior marking was made on both sides of the LIMA and its veins with bi-polar technique. Hereafter the LIMA and its veins were dissected free with scissor and forceps. Clips were added to all side branches. When the full length of LIMA was obtained, the LIMA and its veins were divided distally by adding clips on the peripheral part of the vessels and proximately dividing by scissor. A vessel-clamp was placed distally and the pedicled LIMA placed in the jugular cavity with a cloth containing papaverine.
  Arms: Pedicled
Procedure: Surgical skeletonised — Surgical procedure: The fascia of the LIMA was opened with a scissor. Hereafter the LIMA was dissected free with scissor and forceps, clips on all LIMA side-branches and divided by scissor. When the full length of LIMA was obtained, the LIMA was divided distally by adding clips on the peripheral part of the vessel and proximately dividing by scissor. A vessel-clamp was placed distally, and the skeletonised LIMA placed in the jugular cavity with a cloth containing papaverine.
  Arms: Surgical skeletonised
Procedure: Thunderbeat skeletonised — Surgical procedure: With Thunderbeat the fascia of LIMA was opened. The LIMA was dissected free with Thunderbeat including all side-branches. When the full length of the LIMA was obtained, the LIMA was divided distally by adding clips on the peripheral part of the vessel and proximately dividing by scissor. A vessel-clamp was placed distally, and the skeletonised LIMA placed in the jugular cavity with a cloth containing papaverine.
  Arms: Skeletonised with Thunderbeat

SUMMARY:
It is to date unknown whether Thunderbeat has a place in harvesting the left internal mammary artery (LIMA) and whether skeletonisation is superior to pedicle harvested LIMA. Though, some studies have shown improved flow-rates in the skeletonised graft while others shows compromised blood flow to the thoracic wall after pedicle harvested LIMA.

The purpose of this study is to improve the quality of life for patients undergoing coronary artery bypass graft (CABG) operations.

The aim of this study is to compare three groups of LIMA harvesting techniques: Pedicled, surgical skeletonised and skeletonised with Thunderbeat to determine the best way to harvest LIMA during CABG operations.

The study design is an experimental randomized controlled trial in a single centre.

Study population: Adult patients enlisted for elective stand-alone CABG surgery at the Department of Cardiothoracic surgery, Odense University Hospital.

Study Unit: Test-days within subject and subject

The study will address two main hypotheses in CABG patients:

1. That both the surgical skeletonised and Thunderbeat skeletonised harvesting techniques of LIMA are superior to pedicled harvesting in regards to flowrates and pulsatility index (PI).
2. Skeletonized harvesting of LIMA graft compared to pedicled harvesting improves patient quality of life three days, 30 days, and six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Stand-alone CABG (surgical removal of the left atrial appendage (LAAX) is accepted, since it doesn't affect the graft area)
* On-pump with cardioplegia (otherwise one cannot be sure of the pressure and perfusion during surgery of the graft)
* Patients aged >18
* Elective surgery (there is a known higher risk of postoperative complications with urgent surgery)

Exclusion Criteria:

* CABG combined with other heart surgery, except from LAAX
* Previous heart surgery
* LVEF < 40% (there is a known higher risk of postoperative complications with low LVEF)
* Known cancers (there is a known higher risk of postoperative complication)
* Thoracic radiation therapy (there is a known higher risk of postoperative complication)
* Severe chronic obstructive pulmonary disease (COPD) (there is a known higher risk of postoperative complication)
* Patients not able to understand written consent
* Urgent and emergent surgery (there is a known higher risk of postoperative complication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Differences in flow in LIMA and pulssatility index between the three groups. | Perioperative - After weaning off the extracorporeal circulation just before closing the thorax
  mL/ min With transit time flowmetry (Sono TT flowlab), the graft flow and peripheral index (PI) are measured after weaning off the extracorporeal circulation with a systolic pressure aimed at 100 mmHg. The measurements are done with probe size 3 or 4.

SECONDARY OUTCOMES:
Postoperative bleeding | Postoperative bleeding is measured from the end of the operation to removal of the mediastinal drains in the intensive care unit
  Unit: mL
Re-operation due to bleeding | Up to 48 hours calculated from the end of primaery surgery
  Number of patients in each group
Re-operation due to ischemia | Up to 48 hours calculated from the end of primaery surgery
  Number of patients in each group
Pleurocentesis | Up to 10 days calculated from the end of primaery surgery
  Number of patients in each group
Myocardial injury - creatine kinase-MB (CK-MB) | Routine bloodsample measured four hours after aortic cross clamp removal.
  Unit: (µg/L)
Myocardial injury - cardiac troponin (cTn) | Routine bloodsample measured four hours after aortic cross clamp removal.
  Unit: (ng/L)
Differences in pre and post operative regional oxygen saturation on the thorax. | Measured 7 days prior to surgery and again 3 days after surgery
  Unit: oxygen saturation (rSO2)
Length of stay on ICU | Day of surgery to the day of discharge from ICU. Up to 52 weeks
  Unit: Days
Length of stay in hospital | Day of surgery to the day of discharge from hospital. Up to 52 weeks
  Unit: Days
EQ-5D-5L questionnaire: differences in self reported assessment of patient quality of life between the 3 groups | Questionnaires uptained the week before the date of surgery and again 3, 30, and 180 days after surgery.
  Developed by the EURO-QoF group in 1990 to describe five dimensions of quality of life: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems and a visual analogue scale recording the patient's self-rated health.
Telephone interview - Questions regarding pain, numbness and wound healing around the thoracic incision. | 180 ± 7 days calculated from the date of surgery.
  All questions are closed questions and qualitative variables (yes/no)
Rate of readmission to hospital due to Major adverse cardiac and cerebrovascular events (MACCE) - early | Early (≤30 days)
  Number of deaths in each group
Rate of readmission to hospital due to Major adverse cardiac and cerebrovascular events (MACCE) - Intermediate | Intermediate (≤180 days)
  Number of deaths in each group
Rate of readmission to hospital due to Major adverse cardiac and cerebrovascular events (MACCE) - Long | Long (≤2 years)
  Number of deaths in each group
Rate of mortality due to cardiac event - Early | Early (≤30 days)
  Number of deaths in each group
Rate of mortality due to cardiac event - Intermediate | Intermediate (≤180 days)
  Number of deaths in each group
Rate of mortality due to cardiac event - Iong | Long (≤2 years)
  Number of deaths in each group
Rate of all-cause mortality - Early | Early (≤30 days)
  Number of deaths in each group
Rate of all-cause mortality - Intermediate | Intermediate (≤180 days)
  Number of deaths in each group
Rate of all-cause mortality - long | Long (≤ 2 years)
  Number of deaths in each group

CONTACTS AND LOCATIONS:
Overall Officials: Lars P Riber, MD, Ph.D. DMSc, Study Director — Odense University Hospital
Locations (1):
- Department of Cardio, Vascular and Thoracic Surgery, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Melly L, Torregrossa G, Lee T, Jansens JL, Puskas JD. Fifty years of coronary artery bypass grafting. J Thorac Dis. 2018 Mar;10(3):1960-1967. doi: 10.21037/jtd.2018.02.43. PMID 29707352
- [Background] Thuijs DJFM, Kappetein AP, Serruys PW, Mohr FW, Morice MC, Mack MJ, Holmes DR Jr, Curzen N, Davierwala P, Noack T, Milojevic M, Dawkins KD, da Costa BR, Juni P, Head SJ; SYNTAX Extended Survival Investigators. Percutaneous coronary intervention versus coronary artery bypass grafting in patients with three-vessel or left main coronary artery disease: 10-year follow-up of the multicentre randomised controlled SYNTAX trial. Lancet. 2019 Oct 12;394(10206):1325-1334. doi: 10.1016/S0140-6736(19)31997-X. Epub 2019 Sep 2. PMID 31488373
- [Background] Harskamp RE, Lopes RD, Baisden CE, de Winter RJ, Alexander JH. Saphenous vein graft failure after coronary artery bypass surgery: pathophysiology, management, and future directions. Ann Surg. 2013 May;257(5):824-33. doi: 10.1097/SLA.0b013e318288c38d. PMID 23574989
- [Background] Loop FD, Lytle BW, Cosgrove DM, Stewart RW, Goormastic M, Williams GW, Golding LA, Gill CC, Taylor PC, Sheldon WC, et al. Influence of the internal-mammary-artery graft on 10-year survival and other cardiac events. N Engl J Med. 1986 Jan 2;314(1):1-6. doi: 10.1056/NEJM198601023140101. PMID 3484393
- [Background] Sa MP, Cavalcanti PE, Santos HJ, Soares AF, Miranda RG, Araujo ML, Lima RC. Flow capacity of skeletonized versus pedicled internal thoracic artery in coronary artery bypass graft surgery: systematic review, meta-analysis and meta-regression. Eur J Cardiothorac Surg. 2015 Jul;48(1):25-31. doi: 10.1093/ejcts/ezu344. Epub 2014 Sep 15. PMID 25228742
- [Background] Kamiya H, Akhyari P, Martens A, Karck M, Haverich A, Lichtenberg A. Sternal microcirculation after skeletonized versus pedicled harvesting of the internal thoracic artery: a randomized study. J Thorac Cardiovasc Surg. 2008 Jan;135(1):32-7. doi: 10.1016/j.jtcvs.2007.09.004. PMID 18179915
- [Background] Markman PL, Rowland MA, Leong JY, Van Der Merwe J, Storey E, Marasco S, Negri J, Bailey M, Rosenfeldt FL. Skeletonized internal thoracic artery harvesting reduces chest wall dysesthesia after coronary bypass surgery. J Thorac Cardiovasc Surg. 2010 Mar;139(3):674-9. doi: 10.1016/j.jtcvs.2009.03.066. Epub 2009 Sep 22. PMID 19775705
- [Background] Cheng K, Rehman SM, Taggart DP. A Review of Differing Techniques of Mammary Artery Harvesting on Sternal Perfusion: Time for a Randomized Study? Ann Thorac Surg. 2015 Nov;100(5):1942-53. doi: 10.1016/j.athoracsur.2015.06.087. Epub 2015 Sep 26. PMID 26410160
- [Background] Raja SG, Dreyfus GD. Internal thoracic artery: to skeletonize or not to skeletonize? Ann Thorac Surg. 2005 May;79(5):1805-11. doi: 10.1016/j.athoracsur.2004.05.053. PMID 15854993
- [Background] Lamy A, Browne A, Sheth T, Zheng Z, Dagenais F, Noiseux N, Chen X, Bakaeen FG, Brtko M, Stevens LM, Alboom M, Lee SF, Copland I, Salim Y, Eikelboom J; COMPASS Investigators. Skeletonized vs Pedicled Internal Mammary Artery Graft Harvesting in Coronary Artery Bypass Surgery: A Post Hoc Analysis From the COMPASS Trial. JAMA Cardiol. 2021 Sep 1;6(9):1042-1049. doi: 10.1001/jamacardio.2021.1686. PMID 34132753
- [Background] Liberman M, Khereba M, Goudie E, Kazakov J, Thiffault V, Lafontaine E, Ferraro P. Pilot study of pulmonary arterial branch sealing using energy devices in an ex vivo model. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3219-23. doi: 10.1016/j.jtcvs.2014.05.089. Epub 2014 Jul 19. PMID 25125207
- [Background] Lee SW, Jo JY, Kim WJ, Choi DK, Choi IC. Patient and haemodynamic factors affecting intraoperative graft flow during coronary artery bypass grafting: an observational pilot study. Sci Rep. 2020 Jul 31;10(1):12968. doi: 10.1038/s41598-020-69924-w. PMID 32737380
- [Background] Takami Y, Ina H. Effects of skeletonization on intraoperative flow and anastomosis diameter of internal thoracic arteries in coronary artery bypass grafting. Ann Thorac Surg. 2002 May;73(5):1441-5. doi: 10.1016/s0003-4975(02)03501-4. PMID 12022530
- [Background] Mannacio V, Di Tommaso L, De Amicis V, Stassano P, Vosa C. Randomized flow capacity comparison of skeletonized and pedicled left internal mammary artery. Ann Thorac Surg. 2011 Jan;91(1):24-30. doi: 10.1016/j.athoracsur.2010.06.131. PMID 21172479
- [Background] Mazur P, Litwinowicz R, Tchantchaleishvili V, Natorska J, Zabczyk M, Bochenek M, Przybylski R, Iwaniec T, Kedziora A, Filip G, Kapelak B. Left Internal Mammary Artery Skeletonization Reduces Bleeding-A Randomized Controlled Trial. Ann Thorac Surg. 2021 Sep;112(3):794-801. doi: 10.1016/j.athoracsur.2020.10.024. Epub 2020 Nov 7. PMID 33171172
- [Background] Ben-Yehuda O, Chen S, Redfors B, McAndrew T, Crowley A, Kosmidou I, Kandzari DE, Puskas JD, Morice MC, Taggart DP, Leon MB, Lembo NJ, Brown WM, Simonton CA, Dressler O, Kappetein AP, Sabik JF, Serruys PW, Stone GW. Impact of large periprocedural myocardial infarction on mortality after percutaneous coronary intervention and coronary artery bypass grafting for left main disease: an analysis from the EXCEL trial. Eur Heart J. 2019 Jun 21;40(24):1930-1941. doi: 10.1093/eurheartj/ehz113. PMID 30919909
- [Background] Gahl B, Gober V, Odutayo A, Tevaearai Stahel HT, da Costa BR, Jakob SM, Fiedler GM, Chan O, Carrel TP, Juni P. Prognostic Value of Early Postoperative Troponin T in Patients Undergoing Coronary Artery Bypass Grafting. J Am Heart Assoc. 2018 Feb 27;7(5):e007743. doi: 10.1161/JAHA.117.007743. PMID 29487111
- [Background] Boczor S, Daubmann A, Eisele M, Blozik E, Scherer M. Quality of life assessment in patients with heart failure: validity of the German version of the generic EQ-5D-5L. BMC Public Health. 2019 Nov 6;19(1):1464. doi: 10.1186/s12889-019-7623-2. PMID 31694584
- [Derived] Laugesen S, Krasniqi L, Benhassen LL, Mortensen PE, Pallesen PA, Bak S, Kjelsen BJ, Riber LP. How to harvest the left internal mammary artery-a randomized controlled trial. Interdiscip Cardiovasc Thorac Surg. 2024 May 2;38(5):ivae102. doi: 10.1093/icvts/ivae102. PMID 38775645